CLINICAL TRIAL: NCT06988371
Title: Responses of Adults Smoking Nondaily and Daily in the Experimental Tobacco Marketplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bethany Shorey Fennell (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Bethany Shorey Fennell, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 99596; 5U54DA058256-02 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use; Cigarette Use
Keywords: tobacco; cigarettes; nondaily smoking; behavioral economics
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Mixed crossover-factorial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily smoking (Experimental): Participants who smoke cigarettes every day
  Interventions: Behavioral: Reduced nicotine regulatory environment; Behavioral: Restriction on characterizing flavors in combustible nicotine products; Behavioral: Restriction on characterizing flavors in noncombustible nicotine products
- Nondaily smoking (Experimental): Participants who smoke cigarettes some days but not every day in a month
  Interventions: Behavioral: Reduced nicotine regulatory environment; Behavioral: Restriction on characterizing flavors in combustible nicotine products; Behavioral: Restriction on characterizing flavors in noncombustible nicotine products

INTERVENTIONS:
Behavioral: Reduced nicotine regulatory environment — In this regulatory environment, participants' usual combustible cigarette will not be available in the Experimental Tobacco Marketplace and reduced nicotine content cigarettes will be the only available combustible cigarette.
Behavioral: Restriction on characterizing flavors in combustible nicotine products — In this regulatory environment, menthol and other characterizing flavors in combustible nicotine products will not be available in the Experimental Tobacco Marketplace. Tobacco- or no-flavored combustible nicotine products will be the only combustible nicotine products available.
Behavioral: Restriction on characterizing flavors in noncombustible nicotine products — In this regulatory environment, menthol and other characterizing flavors in noncombustible nicotine products will not be available in the Experimental Tobacco Marketplace. Tobacco- or no-flavored noncombustible nicotine products will be the only noncombustible nicotine products available.

SUMMARY:
The goal of this project is to learn about the potential impact of tobacco regulations that could affect the availability of tobacco products among adults who smoke nondaily and daily. Nondaily smoking is increasingly common and tobacco regulation research should consider how FDA actions may impact this group. Participants will be asked to complete online surveys and tests, online shopping sessions in a simulated Experimental Tobacco Marketplace. Reactions and decisions of adults who smoke nondaily and daily will be compared.

DETAILED DESCRIPTION:
After granting informed consent, participants will complete the single assessment.

First, investigators will collect information from participants on personal characteristics, substance use patterns and addiction severity, and behavioral and cognitive tasks that measure components of our behavioral economic model of product valuation.

Experimental Tobacco Marketplace. In this procedure, participants will complete purchasing scenarios in a realistic tobacco/nicotine product marketplace to model and examine the impact of each of the proposed tobacco product regulations. Participants will be seated in front of a computer to access a simulated online tobacco marketplace with an interface similar to many online merchants. This will allow participants to browse through the selection of tobacco products and add as many as they desire of each product to the virtual shopping cart. Each product will have the price clearly displayed along with an image and description of the product. The selection of products will vary based on the particular regulatory scenario that is being modeled. In each pricing scenario during each marketplace session, participants will be asked to make nicotine-product purchases sufficient for one week's use from this marketplace. During a purchasing session, the participant will be provided with a virtual budget that matches their actual weekly budget for nicotine/tobacco products, a procedure our team has shown to generate realistic results. Participants will use that virtual budget to indicate which selection of products they would purchase from those available in the marketplace.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Consume cigarettes 4-30 days per month
* Have no plans to quit nicotine/tobacco products
* Read and understand English

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Aggregate behavioral economic demand across all participants under the proposed regulatory environments | Baseline
  Participants will complete trials of the Experimental Tobacco Marketplace wherein the price of a target commodity will be increased. Nonlinear mixed effects modeling will be used to fit a curve to estimate the number of products purchased at each price and the analysis will result in an measure of overall price sensitivity under each of the regulatory conditions.
Aggregate behavioral economic substitution across all participants under the proposed regulatory environments | Baseline
  Participants will complete trials of the Experimental Tobacco Marketplace wherein the price of alternative products will be fixed across trials and their usual product will change price. Mixed effects modeling will be used to fit a curve to estimate the slopes and intercepts of these alternative products, revealing the degree to which participants will choose to purchase each alternative product as the price of the participant's usual product increases.

SECONDARY OUTCOMES:
Hypothetical quantity purchased in purchase tasks | Baseline
  Measures valuation by assessing hypothetical consumption across a price range and across the range of products used by participants in the past 60 days.
Delay Discounting Tasks | Baseline
  Assesses valuation for future money and nicotine products.

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Shorey Fennell, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified data will be shared.

DOCUMENTS (1):
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT06988371/ICF_000.pdf